CLINICAL TRIAL: NCT00804882
Title: Correlation in Hispanics of Accelerated Metabolic Risk Profile and Non-ischemic Heart Failure (CHAMP-HF)
Brief Title: Hispanics With Metabolic Syndrome and Non-ischemic Heart Failure
Acronym: CHAMP-HF
Status: Withdrawn | Type: Observational
Why Stopped: Principal investigator is leaving the institution to obtain further training.
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Rey Vivo, MD, Texas Tech University Health Sciences Center
Other Study IDs: L08-174
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Metabolic Syndrome; Heart Failure
Keywords: Metabolic syndrome; Heart failure; Mexican Americans; Ethnic differences; Echocardiography
MeSH Terms: conditions — Metabolic Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Mexican Americans with heart failure and metabolic syndrome
- 2: Mexican Americans with heart failure without metabolic syndrome
- 3: Non-Hispanic White Americans with heart failure and metabolic syndrome
- 4: Non-Hispanic White Americans with heart failure without metabolic syndrome

SUMMARY:
The investigators aim to examine how medical conditions that indicate high cardiometabolic risk, such as increased body weight, high cholesterol levels and high blood pressure, affect heart structure and function among individuals with known HF. Furthermore, this study is being undertaken to identify potential differences in these effects between non-Hispanics whites and Mexican Americans.

DETAILED DESCRIPTION:
While it is known that Mexican Americans are inordinately affected by metabolic syndrome (MetS), it is unclear how metabolic risk factors impact left ventricular structure and function in Mexican Americans with HF. There is also a gap in the knowledge of the principal etiology of HF in this ethnic group. The overall objective of this pilot study is to define the association between MetS and and non-ischemic HF in Mexican Americans. Our central hypothesis is that there is a positive graded association between an increasing number of metabolic risk factors (ie. individual components of MetS) and increasingly compromised LV structure and function in this population, independent of blood pressure and CAD. Additionally, we hypothesize that this association is more pronounced than that seen in non-Hispanic whites suggesting a predominant role of MetS on HF among Mexican Americans. The rationale that underlies the proposed research is that, once the association between metabolic risk factors and HF in this ethnic group is defined, future research on the impact of management of these metabolic risk factors on HF outcomes, both among Mexican Americans and in the larger population, will be advanced.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-59 years
2. known diagnosis of HF
3. complete 2-dimensional and Doppler echocardiogram within the last 12 months.

Exclusion Criteria:

1. history of CAD determined by recorded or self-reported history of CAD and/or revascularization
2. recent history (previous 6 months) of decompensated HF
3. heart transplant
4. diagnosis of diabetes (rationale: diabetes independently predicts HF)
5. race/ethnicity other than Mexican American or non-Hispanic white.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mexican Americans and Non-Hispanic White Americans with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Evaluate ethnicity-specific differences in the association between increasing number of metabolic risk factors and increasingly compromised LV structure and function among Mexican Americans, in comparison to non-Hispanic whites. | Within 1 week of enrollment

SECONDARY OUTCOMES:
Compare the severity of MetS between a cross-sectional sample of Mexican American adults and an age- and gender-matched population of non-Hispanic whites with an established diagnosis of non-ischemic HF | Within one week of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Rey P Vivo, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States